CLINICAL TRIAL: NCT05429151
Title: Clinical and Dermoscopic Study of Intralesional Injection of Acyclovir Versus Candida Antigen in Treatment of Plantar Warts
Brief Title: Intralesional Injection of Acyclovir Versus Candida Antigen in Treatment of Plantar Warts
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Raghda Mohamed Hassan, resident at dermatology venereology andrology department, Sohag University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-22-06-06
Record Dates: First submitted 2022-06-13; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Acyclovir and Candida Antigen in Treatment of Plantar Wart
Keywords: acyclovir ,candida antigen ,plantar wart
MeSH Terms: interventions — Acyclovir; Powders; Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): will be treated with intralesional injection of acyclovir (Acyclovir 250mg Powder for Solution for Infusion, each vial contains 250mg of acyclovir as the sodium salt, Chandra Bhagat Pharma Pvt. Ltd) 250 mg acyclovir vial diluted with 3.5 ml saline to get approximately 70 mg/ml solution. During the study, the dosage of the drug and frequency of treatment were uniform in all patients. The base of each wart was injected with 0.1 ml of intralesional acyclovir (70 mg/ml) using an insulin syringe (29 Gage × 0.5-in) every 2 weeks until the resolution of warts or for a maximum of 5 sessions
  Interventions: Drug: Acyclovir 250mg Powder for Solution for Infusion, each vial contains 250mg of acyclovir as the sodium salt, Chandra Bhagat Pharma Pvt. Ltd andcandida antigen
- group 2 (Active Comparator): will be treated by intralesional Candida antigen injection (candida antigen ) at a dose of 0.2 mL. injected into the largest wart using an insulin syringe (29 Gage × 0.5-in) every 2 weeks until complete clearance of warts or for a maximum of 5 treatment sessions.
  Interventions: Drug: Acyclovir 250mg Powder for Solution for Infusion, each vial contains 250mg of acyclovir as the sodium salt, Chandra Bhagat Pharma Pvt. Ltd andcandida antigen

INTERVENTIONS:
Drug: Acyclovir 250mg Powder for Solution for Infusion, each vial contains 250mg of acyclovir as the sodium salt, Chandra Bhagat Pharma Pvt. Ltd andcandida antigen — Group 1: will be treated with intralesional injection of acyclovir (Acyclovir 250mg Powder for Solution for Infusion, each vial contains 250mg of acyclovir as the sodium salt, Chandra Bhagat Pharma Pvt. Ltd) 250 mg acyclovir vial diluted with 3.5 ml saline to get approximately 70 mg/ml solution. During the study, the dosage of the drug and frequency of treatment were uniform in all patients. The base of each wart was injected with 0.1 ml of intralesional acyclovir (70 mg/ml) using an insulin syringe (29 Gage × 0.5-in) every 2 weeks until the resolution of warts or for a maximum of 5 sessions
  Group 2: will be treated by intralesional Candida antigen injection (candida antigen ) at a dose of 0.2 mL. injected into the largest wart using an insulin syringe (29 Gage × 0.5-in) every 2 weeks until complete clearance of warts or for a maximum of 5 treatment sessions.

SUMMARY:
This study aims to evaluate the efficacy of intralesional injection of acyclovir versus candida antigen in plantar wart patients will be randomly divided into 2 groups,At least 20 patients will be enrolled in each group.

Group 1: will be treated with intralesional injection of acyclovir 250 mg acyclovir vial diluted with 3.5 ml saline to get approximately 70 mg/ml solution. The base of each wart was injected with 0.1 ml of intralesional acyclovir (70 mg/ml) every 2 weeks until the resolution of warts or for a maximum of 5 sessions Group 2: will be treated by intralesional Candida antigen injection (candida antigen ) at a dose of 0.2 mL. injected into the largest wart every 2 weeks until complete clearance of warts or for a maximum of 5 treatment sessions.

3.Patient evaluation: Assessment of treatment efficacy and side effects will be carried out by clinical examination and comparative photographic evaluation and dermoscopy

DETAILED DESCRIPTION:
patients will be randomly divided into 2 groups, group (1) and group (2). At least 20 patients will be enrolled in each group.

Group 1: will be treated with intralesional injection of acyclovir (Acyclovir 250mg Powder for Solution for Infusion, each vial contains 250mg of acyclovir as the sodium salt, Chandra Bhagat Pharma Pvt. Ltd) 250 mg acyclovir vial diluted with 3.5 ml saline to get approximately 70 mg/ml solution. During the study, the dosage of the drug and frequency of treatment were uniform in all patients. The base of each wart was injected with 0.1 ml of intralesional acyclovir (70 mg/ml) using an insulin syringe (29 Gage × 0.5-in) every 2 weeks until the resolution of warts or for a maximum of 5 sessions

Group 2: will be treated by intralesional Candida antigen injection (candida antigen ) at a dose of 0.2 mL. injected into the largest wart using an insulin syringe (29 Gage × 0.5-in) every 2 weeks until complete clearance of warts or for a maximum of 5 treatment sessions.

patients will be followed up for 3months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with single or multiple planter wart. Age group 18:50 years old

Exclusion Criteria:

* : patients with history of renal or liver disease, pregnant and lactating females, patients taking immunosuppressant drugs, patients who received any treatment for wart in the last month before the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
degree of improvment of wart after intralesional injection of acyclovir and candida antigen | 3months after treatment.
  1. complete response: when 100% complete disappearance of the wart.
  2. partial response: if there is 50% to 99% reduction in its original diameter.
  3. no response: if there reduction in its size <50% .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No